CLINICAL TRIAL: NCT02525939
Title: A Phase III, Double-blind, Randomized Placebo-controlled Study to Evaluate the Effects of Dalcetrapib on Cardiovascular (CV) Risk in a Genetically Defined Population With a Recent Acute Coronary Syndrome (ACS): The Dal-GenE Trial
Brief Title: Effect of Dalcetrapib vs Placebo on CV Risk in a Genetically Defined Population With a Recent ACS
Acronym: dal-GenE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: DalCor Pharmaceuticals (Industry)
Collaborators: The Montreal Health Innovations Coordinating Center (MHICC) (Other); Medpace, Inc. (Industry); Roche Molecular Systems, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAL-301
Record Dates: First submitted 2015-08-13; First posted 2015-08-18 (Estimated); Results first posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-09

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — dalcetrapib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dalcetrapib (Active Comparator): Participants received dalcetrapib 600 mg (two 300 mg tablets) orally once daily.
  dalcetrapib: Cholesterol Ester Transfer Protein inhibitor, 300 mg tablets
  Interventions: Drug: dalcetrapib
- Placebo (Placebo Comparator): Participants received dalcetrapib placebo tablets matching dalcetrapib orally once daily.
  Placebo: dalcetrapib matching placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: dalcetrapib — Cholesterol Ester Transfer Protein inhibitor
  Arms: Dalcetrapib
Drug: Placebo — matching placebo tablets
  Arms: Placebo

SUMMARY:
A placebo-controlled, randomized, double-blind, parallel group, phase III multicenter study in subjects recently hospitalized for ACS and with the appropriate genetic profile. Subjects will provide informed consent before any study-specific procedures are performed. Subject enrollment may begin in the hospital and will continue following release from the hospital. Screening procedures may be performed at the time of the index ACS event or anytime thereafter, with the condition that randomization must occur within the mandated window (4-12 weeks after the index event). Subjects will be assessed based on their medical history. Those who are likely to qualify will undergo Genotype Assay testing to evaluate genetic determination for the presence of AA genotype.

DETAILED DESCRIPTION:
This is an event driven study to reach statistical power given all other assumptions. Subjects will visit the clinic 1 month after randomization and at regular intervals thereafter. Additionally, for any subject prematurely discontinuing study medication, assessments will be conducted every 6 months for the collection of study endpoints.

Those who are likely to qualify will undergo Genotype Assay Testing to evaluate genetic determination or the presence of the AA genotype. The test is investigational and test procedures are Roche Molecular Diagnostics protocol ADCY9-COB-389.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with the appropriate genetic background and recently hospitalized for ACS (between 4 and 12 weeks following the index event), will be enrolled in this trial.
* AA genotype at variant gene as determined by Genotype Assay testing, conducted at a designated investigational testing site (ITS)
* Clinically stable, ie, free of ischemic symptoms at rest or with minimal exertion for at least 1 week prior to randomization
* Prior to randomization, subject must have evidence of guidelines-based management of LDL-C, at a minimum to include medical and dietary treatment to a target level of LDL-C <100 mg/dl (<2.6 mmol/L).

Exclusion Criteria:

* Females who are pregnant (negative pregnancy test required for all women of child-bearing potential at Visit 2, Day 0) or breast-feeding
* Women of childbearing potential (women who are not surgically sterile or postmenopausal defined as amenorrhea for >12 months) who are not using at least one method of contraception*
* New York Heart Association (NYHA) Class III or IV heart failure
* Last known hemoglobin <10 g/dL
* Index ACS event presumed due to uncontrolled hypertension

(*) Varies by region

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6147 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2021-10 (Actual); Study Completion 2021-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald M Black, MD, Study Director — DalCor Pharmaceuticals
Locations (557):
- United States (122):
  - Research Site, Alexander City, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Cottonwood, Arizona
  - Research Site, Glendale, Arizona
  - Research Site, Jonesboro, Arkansas
  - Research Site, Huntington Beach, California
  - Research Site, San Diego, California
  - Research Site, Torrance, California
  - Research Site, Denver, Colorado
  - Research Site, Littleton, Colorado
  - Research Site, Danbury, Connecticut
  - Research Site, Hartford, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Clearwater, Florida
  - Research Site, Daytona Beach, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Homestead, Florida
  - Research Site, Hudson, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Largo, Florida
  - Research Site, Miami, Florida
  - Research Site, Miramar, Florida
  - Research Site, Orlando, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Safety Harbor, Florida
  - Research Site, Tallahassee, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Covington, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Evanston, Illinois
  - Research Site, Jerseyville, Illinois
  - Research Site, Fort Wayne, Indiana
  - Research Site, Newburgh, Indiana
  - Research Site, West Des Moines, Iowa
  - Research Site, Wichita, Kansas
  - Research Site, Owensboro, Kentucky
  - Research Site, Alexandria, Louisiana
  - Research Site, Covington, Louisiana
  - Research Site, Bangor, Maine
  - Research Site, Biddeford, Maine
  - Research Site, Lewiston, Maine
  - Research Site, Annapolis, Maryland
  - Research Site, Baltimore, Maryland
  - Research Site, Bethesda, Maryland
  - Research Site, Columbia, Maryland
  - Research Site, Salisbury, Maryland
  - Research Site, Hyannis, Massachusetts
  - Research Site, Alpena, Michigan
  - Research Site, Bay City, Michigan
  - Research Site, Lansing, Michigan
  - Research Site, Midland, Michigan
  - Research Site, Mount Clemens, Michigan
  - Research Site, Muskegon, Michigan
  - Research Site, Saginaw, Michigan
  - Research Site, Saint Joseph, Michigan
  - Research Site, Ypsilanti, Michigan
  - Research Site, Coon Rapids, Minnesota
  - Research Site, Duluth, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Saint Cloud, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Washington, Missouri
  - Research Site, Missoula, Montana
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Bridgewater, New Jersey
  - Research Site, Linden, New Jersey
  - Research Site, Somerset, New Jersey
  - Research Site, Summit, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Buffalo, New York
  - Research Site, Johnson City, New York
  - Research Site, New Windsor, New York
  - Research Site, New York, New York
  - Research Site, Poughkeepsie, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Pinehurst, North Carolina
  - Research Site, Rocky Mount, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Minot, North Dakota
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Springfield, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Zanesville, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Butler, Pennsylvania
  - Research Site, Chambersburg, Pennsylvania
  - Research Site, Erie, Pennsylvania
  - Research Site, Hershey, Pennsylvania
  - Research Site, Langhorne, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Wyomissing, Pennsylvania
  - Research Site, York, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Spartanburg, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Greeneville, Tennessee
  - Research Site, Jackson, Tennessee
  - Research Site, Oak Ridge, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Kingwood, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Victoria, Texas
  - Research Site, Wichita Falls, Texas
  - Research Site, Layton, Utah
  - Research Site, Charlottesville, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Virginia Beach, Virginia
  - Research Site, Winchester, Virginia
  - Research Site, Seattle, Washington
  - Research Site, La Crosse, Wisconsin
- Argentina (24):
  - Research Site, Bahía Blanca
  - Research Site, Buenos Aires
  - Research Site, Coronel Suárez
  - Research Site, Corrientes
  - Research Site, Córdoba
  - Research Site, Esperanza
  - Research Site, Junín
  - Research Site, La Plata
  - Research Site, Mar del Plata
  - Research Site, Mendoza
  - Research Site, Morón
  - Research Site, Quilmes
  - Research Site, Rosario
  - Research Site, San Juan
  - Research Site, San Luis
  - Research Site, San Martín
  - Research Site, San Miguel de Tucumán
  - Research Site, San Nicolás
  - Research Site, Santa Fe
  - Research Site, Santa Rosa
  - Research Site, Venado Tuerto
  - Research Site, Vicente López
  - Research Site, Villa Allende
  - Research Site, Villa María
- Australia (22):
  - Research Site, Bruce, New South Wales
  - Research Site, Gosford, New South Wales
  - Research Site, Liverpool, New South Wales
  - Research Site, Saint Leonards, New South Wales
  - Research Site, Cairns, Queensland
  - Research Site, Chermside, Queensland
  - Research Site, Douglas, Queensland
  - Research Site, Herston, Queensland
  - Research Site, Milton, Queensland
  - Research Site, Redcliffe, Queensland
  - Research Site, Woolloongabba, Queensland
  - Research Site, Bedford Park, South Australia
  - Research Site, Elizabeth Vale, South Australia
  - Research Site, Woodville South, South Australia
  - Research Site, Hobart, Tasmania
  - Research Site, Epping, Victoria
  - Research Site, Geelong, Victoria
  - Research Site, Melbourne, Victoria
  - Research Site, Joondalup, Western Australia
  - Research Site, Murdoch, Western Australia
  - Research Site, Nedlands, Western Australia
  - Research Site, Perth, Western Australia
- Austria (6):
  - Research Site, Braunau am Inn
  - Research Site, Feldkirch
  - Research Site, Krems
  - Research Site, Linz
  - Research Site, Vienna
  - Research Site, Wiener Neustadt
- Belgium (9):
  - Research Site, Aalst
  - Research Site, Bonheiden
  - Research Site, Brussels
  - Research Site, Genk
  - Research Site, Liège
  - Research Site, Maaseik
  - Research Site, Mechelen
  - Research Site, Ottignies
  - Research Site, Sint-Niklaas
- Brazil (21):
  - Research Site, Belo Horizonte
  - Research Site, Blumenau
  - Research Site, Brasília
  - Research Site, Campina Grande do Sul
  - Research Site, Campinas
  - Research Site, Campo Grande
  - Research Site, Curitiba
  - Research Site, Fortaleza
  - Research Site, Goiânia
  - Research Site, Maringá
  - Research Site, Marília
  - Research Site, Natal
  - Research Site, Porto Alegre
  - Research Site, Recife
  - Research Site, Ribeirão Preto
  - Research Site, Salvador
  - Research Site, Santo André
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
  - Research Site, Uberlândia
  - Research Site, Vitória
- Bulgaria (9):
  - Research Site, Blagoevgrad
  - Research Site, Dimitrovgrad
  - Research Site, Haskovo
  - Research Site, Pazardzhik
  - Research Site, Pernik
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Sandanski
  - Research Site, Sofia
- Canada (36):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Moncton, New Brunswick
  - Research Site, Saint John, New Brunswick
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Bridgewater, Nova Scotia
  - Research Site, Burlington, Ontario
  - Research Site, Cambridge, Ontario
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Peterborough, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Thunder Bay, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Granby, Quebec
  - Research Site, Laval, Quebec
  - Research Site, Lévis, Quebec
  - Research Site, Longueuil, Quebec
  - Institut de Cardiologie de Montreal, Montreal, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Saint George, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Saint-Jean-sur-Richelieu, Quebec
  - Research Site, Saint-Jérôme, Quebec
  - Research Site, Sherbrooke, Quebec
  - Research Site, Terrebonne, Quebec
  - Research Site, Thetford-Mines, Quebec
  - Research Site, Trois-Rivières, Quebec
  - Research Site, Québec
- Chile (3):
  - Research Site, Santiago
  - Research Site, Temuco
  - Research Site, Viña del Mar
- Czechia (14):
  - Research Site, Bílina
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Jihlava
  - Research Site, Kladno
  - Research Site, Kroměříž
  - Research Site, Liberec
  - Research Site, Náchod
  - Research Site, Pilsen
  - Research Site, Písek
  - Research Site, Prague
  - Research Site, Slaný
  - Research Site, Trutnov
  - Research Site, Zlín
- Denmark (9):
  - Research Site, Aalborg
  - Research Site, Copenhagen
  - Research Site, Frederiksberg
  - Research Site, Glostrup Municipality
  - Research Site, Hellerup
  - Research Site, Herning
  - Research Site, Hillerød
  - Research Site, Næstved
  - Research Site, Silkeborg
- Finland (4):
  - Research Site, Jyväskylä
  - Research Site, Oulu
  - Research Site, Pori
  - Research Site, Turku
- France (14):
  - Research Site, Besançon
  - Research Site, Bron
  - Research Site, Clermont-Ferrand
  - Research Site, Corbeil-Essonnes
  - Research Site, Dijon
  - Research Site, Limoges
  - Research Site, Lyon
  - Research Site, Montpellier
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Poitiers
  - Research Site, Toulouse
  - Research Site, Tourcoing
  - Research Site, Valenciennes
- Germany (14):
  - Research Site, Aachen
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Bremen
  - Research Site, Chemnitz
  - Research Site, Coburg
  - Research Site, Dresden
  - Research Site, Erfurt
  - Research Site, Fürth
  - Research Site, Heidelberg
  - Research Site, Leipzig
  - Research Site, Mainz
  - Research Site, Mönchengladbach
  - Research Site, Munich
- Hungary (13):
  - Research Site, Baja
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Eger
  - Research Site, Gyula
  - Research Site, Hatvan
  - Research Site, Kecskemét
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Székesfehérvár
  - Research Site, Szombathely
  - Research Site, Zalaegerszeg
- Israel (17):
  - Research Site, Afula
  - Research Site, Ashkelon
  - Research Site, Beersheba
  - Research Site, Bnei Brak
  - Research Site, Haifa
  - Research Site, Holon
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Nahariya
  - Research Site, Nazareth
  - Research Site, Petah Tikva
  - Research Site, Poria Illit
  - Research Site, Rehovot
  - Research Site, Safed
  - Research Site, Tel Aviv
  - Research Site, Tel Litwinsky
  - Research Site, Ẕerifin
- Italy (21):
  - Research Site, Ancona
  - Research Site, Ascoli Piceno
  - Research Site, Cagliari
  - Research Site, Casarano
  - Research Site, Cortona
  - Research Site, Empoli
  - Research Site, Florence
  - Research Site, Foggia
  - Research Site, Giugliano in Campania
  - Research Site, Gubbio
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Novara
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, Sanremo
  - Research Site, Saronno
  - Research Site, Scorrano
  - Research Site, Seriate
  - Research Site, Torino
  - Research Site, Treviglio
- Netherlands (24):
  - Research Site, 's-Hertogenbosch
  - Research Site, Amsterdam
  - Research Site, Arnhem
  - Research Site, Capelle aan den IJssel
  - Research Site, Deventer
  - Research Site, Doetinchem
  - Research Site, Ede
  - Research Site, Goes
  - Research Site, Gouda
  - Research Site, Hoogeveen
  - Research Site, Hoorn
  - Research Site, Leeuwarden
  - Research Site, Leiden
  - Research Site, Rotterdam
  - Research Site, Schiedam
  - Research Site, Sneek
  - Research Site, The Hague
  - Research Site, Tiel
  - Research Site, Tilburg
  - Research Site, Uden
  - Research Site, Veldhoven
  - Research Site, Venlo
  - Research Site, Zaandam
  - Research Site, Zutphen
- New Zealand (11):
  - Research Site, Christchurch
  - Research Site, Dunedin
  - Research Site, Grafton
  - Research Site, Hamilton
  - Research Site, Hastings
  - Research Site, Lower Hutt
  - Research Site, Nelson
  - Research Site, New Plymouth
  - Research Site, Rotorua
  - Research Site, Takapuna
  - Research Site, Wellington
- Poland (20):
  - Research Site, Bydgoszcz
  - Research Site, Elblag
  - Research Site, Gdynia
  - Research Site, Kielce
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Mrągowo
  - Research Site, Oświęcim
  - Research Site, Oława
  - Research Site, Poznan
  - Research Site, Płock
  - Research Site, Ruda Śląska
  - Research Site, Rzeszów
  - Research Site, Sopot
  - Research Site, Szczecin
  - Research Site, Środa Wielkopolska
  - Research Site, Torun
  - Research Site, Wroclaw
  - Research Site, Zabrze
  - Research Site, Zamość
- Portugal (8):
  - Research Site, Almada
  - Research Site, Braga
  - Research Site, Coimbra
  - Research Site, Faro
  - Research Site, Leiria
  - Research Site, Lisbon
  - Research Site, Senhora da Hora
  - Research Site, Setúbal
- Puerto Rico (3):
  - Research Site, Bayamón
  - Research Site, Caguas
  - Research Site, Ponce
- Romania (10):
  - Research Site, Arad
  - Research Site, Baia Mare
  - Research Site, Brăila
  - Research Site, Bucharest
  - Research Site, Buzău
  - Research Site, Cluj-Napoca
  - Research Site, Craiova
  - Research Site, Oradea
  - Research Site, Piteşti
  - Research Site, Timișoara
- Russia (20):
  - Research Site, Arkhangelsk
  - Research Site, Barnaul
  - Research Site, Irkutsk
  - Research Site, Kazan'
  - Research Site, Kemerovo
  - Research Site, Kirovsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Orenburg
  - Research Site, Penza
  - Research Site, Petrozavodsk
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Tomsk
  - Research Site, Tula
  - Research Site, Tyumen
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
- Slovakia (6):
  - Research Site, Bardejov
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Lučenec
  - Research Site, Námestovo
  - Research Site, Nitra
- South Africa (9):
  - Research Site, Bloemfontein
  - Research Site, Cape Town
  - Research Site, Gatong
  - Research Site, Johannesburg
  - Research Site, Kuils River
  - Research Site, Paarl
  - Research Site, Parow
  - Research Site, Somerset West
  - Research Site, Worcester
- Spain (14):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Hospitalet Del Llobregat
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Sabadell
  - Research Site, Salamanca
  - Research Site, Sant Joan
  - Research Site, Santiago de Compostela
  - Research Site, Seville
  - Research Site, Tarragona
  - Research Site, Valencia
  - Research Site, Vigo
- Sweden (9):
  - Research Site, Falun
  - Research Site, Karlshamn
  - Research Site, Köping
  - Research Site, Linköping
  - Research Site, Malmo
  - Research Site, Örebro
  - Research Site, Umeå
  - Research Site, Uppsala
  - Research Site, Västerås
- Switzerland (2):
  - Research Site, Geneva
  - Research Site, Lugano
- Turkey (Türkiye) (9):
  - Research Site, Afyonkarahisar
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Kadıköy
  - Research Site, Kayseri
  - Research Site, Mersin
  - Research Site, Samsun
  - Research Site, Sivas
- United Arab Emirates (2):
  - Research Site, Dubai
  - Research Site, Sharjah city
- United Kingdom (52):
  - Research Site, Ayr
  - Research Site, Barnet
  - Research Site, Basildon
  - Research Site, Belfast
  - Research Site, Birmingham
  - Research Site, Blackpool
  - Research Site, Bradford
  - Research Site, Bristol
  - Research Site, Burton-on-Trent
  - Research Site, Chelmsford
  - Research Site, Chertsey
  - Research Site, Clydebank
  - Research Site, Coventry
  - Research Site, Craigavon
  - Research Site, Dartford
  - Research Site, Dudley
  - Research Site, Glasgow
  - Research Site, Harrow
  - Research Site, High Wycombe
  - Research Site, Hull
  - Research Site, Inverness
  - Research Site, Kirkcaldy
  - Research Site, Lanark
  - Research Site, Leicester
  - Research Site, Lincoln
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Londonderry
  - Research Site, Luton
  - Research Site, Manchester
  - Research Site, Newcastle
  - Research Site, Newport
  - Research Site, Northampton
  - Research Site, Nuneaton
  - Research Site, Paisley
  - Research Site, Redhill
  - Research Site, Romford
  - Research Site, Rotherham
  - Research Site, Salford
  - Research Site, Sheffield
  - Research Site, Stevenage
  - Research Site, Stockport
  - Research Site, Stockton-on-Tees
  - Research Site, Swindon
  - Research Site, Taunton
  - Research Site, Telford
  - Research Site, Truro
  - Research Site, West Bromwich
  - Research Site, Westcliff-on-Sea
  - Research Site, Wigan
  - Research Site, Worcester
  - Research Site, Worthing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tardif JC, Pfeffer MA, Kouz S, Koenig W, Maggioni AP, McMurray JJV, Mooser V, Waters DD, Gregoire JC, L'Allier PL, Wouter Jukema J, White HD, Heinonen T, Black DM, Laghrissi-Thode F, Levesque S, Guertin MC, Dube MP; dal-GenE Investigators. Pharmacogenetics-guided dalcetrapib therapy after an acute coronary syndrome: the dal-GenE trial. Eur Heart J. 2022 Oct 14;43(39):3947-3956. doi: 10.1093/eurheartj/ehac374. PMID 35856777
- [Derived] Black DM, Miller M, Heinonen TM, Zhang G. Advancing Beyond Failed High-density Lipoprotein Clinical Trials to Pharmacogenetic Studies of ADCY9 and Cholesterol Ester Transfer Protein Inhibition. J Cardiovasc Pharmacol. 2021 Oct 1;78(4):496-500. doi: 10.1097/FJC.0000000000001093. PMID 34173811
- [Derived] Tardif JC, Dube MP, Pfeffer MA, Waters DD, Koenig W, Maggioni AP, McMurray JJV, Mooser V, White HD, Heinonen T, Black DM, Guertin MC; dal-GenE Investigators. Study design of Dal-GenE, a pharmacogenetic trial targeting reduction of cardiovascular events with dalcetrapib. Am Heart J. 2020 Apr;222:157-165. doi: 10.1016/j.ahj.2020.01.007. Epub 2020 Jan 17. PMID 32087417

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial enrolment began in April 2016 and was completed in December 2018. A total of 45,005 patients with recent acute coronary syndrome were screened in order to identify participants meeting the single genetic criterion (AA genotype at rs1967309 in the ADCY9 gene) and other inclusion criteria and no exclusion criteria required for randomization.
Pre-assignment Details: A total of 6149 eligible patients underwent randomization, among whom two were randomized by error and excluded.
Period: Overall Study
Arm/Group | Dalcetrapib | Placebo
Started | 3071 | 3076
Took Study Medication | 3064 | 3064
Completed | 2840 | 2833
Not Completed | 231 | 243
Not completed — Lost to Follow-up | 27 | 24
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 24 | 39
Not completed — Death | 180 | 179

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dalcetrapib | Placebo | Total
Number analyzed (Participants) | 3071 | 3076 | 6147
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.19 (9.16) | 62.34 (9.25) | 62.26 (9.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 723 | 672 | 1395
  Male | 2348 | 2404 | 4752
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 469 | 469 | 938
  Not Hispanic or Latino | 2551 | 2550 | 5101
  Unknown or Not Reported | 51 | 57 | 108
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 12 | 23
  Asian | 58 | 59 | 117
  Native Hawaiian or Other Pacific Islander | 15 | 15 | 30
  Black or African American | 130 | 123 | 253
  White | 2771 | 2798 | 5569
  More than one race | 85 | 68 | 153
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United Arab Emirates | 9 | 7 | 16
  Argentina | 74 | 74 | 148
  Australia | 100 | 102 | 202
  Austria | 23 | 27 | 50
  Belgium | 22 | 17 | 39
  Bulgaria | 201 | 185 | 386
  Brazil | 218 | 213 | 431
  Canada | 209 | 228 | 437
  Switzerland | 21 | 15 | 36
  Chile | 44 | 50 | 94
  Czechia | 73 | 78 | 151
  Germany | 28 | 41 | 69
  Denmark | 66 | 71 | 137
  Spain | 84 | 104 | 188
  Finland | 9 | 11 | 20
  France | 49 | 50 | 99
  United Kingdom | 200 | 183 | 383
  Hungary | 82 | 101 | 183
  Israel | 198 | 175 | 373
  Italy | 69 | 54 | 123
  Netherlands | 129 | 147 | 276
  New Zealand | 75 | 74 | 149
  Poland | 166 | 169 | 335
  Puerto Rico | 10 | 4 | 14
  Romania | 92 | 87 | 179
  Russia | 215 | 240 | 455
  Slovakia | 21 | 27 | 48
  Sweden | 35 | 30 | 65
  Turkey | 31 | 26 | 57
  United States | 370 | 358 | 728
  South Africa | 121 | 101 | 222
  Portugal | 27 | 27 | 54
Reproductive status if female [Count of Participants; unit: Participants] — Population: Only female subjects are considered in this baseline measure.
  Participants
    number analyzed (Participants) | 723 | 672 | 1395
    Childbearing potential with double contraceptive protection | 24 | 24 | 48
    Childbearing potential without double contraceptive potential | 1 | 1 | 2
    Postmenopausal | 602 | 584 | 1186
    Surgically sterilized | 92 | 60 | 152
    Other | 4 | 3 | 7
Acute Coronary Syndrome (ACS) Index Event Details: [Mean (Standard Deviation); unit: days]
  Time since ACS index event | 53.82 (18.09) | 54.01 (18.31) | 53.91 (18.20)
  Hospitalization duration | 6.06 (4.33) | 6.22 (5.03) | 6.14 (4.69)
Acute Coronary Syndrome (ACS) Index Event Diagnosis [Count of Participants; unit: Participants]
  Spontaneous Myocardial Infarction (MI) | 2756 | 2742 | 5498
  Procedure-related Myocardial Infarction (MI) after Percutaneous Coronary Intervention (PCI) | 20 | 28 | 48
  Hospitalization for Acute Coronary Syndrome (Electrocardiogram abnormalities without biomarkers) | 295 | 306 | 601
Acute Coronary Syndrome (ACS) Index Event Diagnosis: Second ACS event since qualifying index event [Count of Participants; unit: Participants]
  No | 2998 | 3008 | 6006
  Yes | 73 | 68 | 141

OUTCOME MEASURES:

1. Primary Outcome: Composite of Cardiovascular Death, Resuscitated Cardiac Arrest, Non-Fatal Myocardial Infarction, and Non-Fatal Stroke
Description: All efficacy endpoints were adjudicated by an independent clinical endpoint committee (CEC). The primary efficacy endpoint was the time from randomization to the first occurrence of any component of the composite endpoint, which included death from cardiovascular causes, resuscitated cardiac arrest, non-fatal myocardial infarction, or non-fatal stroke, as positively adjudicated by the CEC.
Time Frame: From randomization to the first occurrence of any component of the composite primary endpoint (median duration of follow-up was 39.9 months)
Population: All subjects randomized to treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dalcetrapib
Number analyzed (Participants) | 3076 | 3071
Participants | 327 | 292
Statistical Analysis 1: Comparison: Placebo vs Dalcetrapib; A stratified Cox proportional hazards model was used to analyze the primary endpoint. This model included treatment as a main effect, and region and acute coronary syndrome (ACS) index event type as stratification factors. The null and alternative hypotheses tested with the above Cox model were: H0: λ = 1 vs HA: λ ≠ 1, where λ is the, assumed constant, hazard ratio (HR) for the time to occurrence of the composite events of the primary endpoint for the dalcetrapib and placebo treated groups; Test type: Superiority; p = 0.12, Stratified Cox proportional hazard model — The estimated HR was presented with a 95% CI and a p-value. The primary analysis was conducted at the 0.05 significance level; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.75 to 1.03]

2. Secondary Outcome: Composite Endpoint of Cardiovascular Death, Resuscitated Cardiac Arrest, Non-Fatal Myocardial Infarction, Non-Fatal Stroke, Hospitalization for ACS (With Electrocardiogram Abnormalities) or Unanticipated Coronary Revascularization
Description: All efficacy endpoints were adjudicated by an independent clinical endpoint committee (CEC). The primary efficacy endpoint was the time from randomization to the first occurrence of any component of the composite endpoint, which included death from cardiovascular causes, resuscitated cardiac arrest, non-fatal myocardial infarction, non-fatal stroke, hospitalization for acute coronary syndrome (with electrocardiogram abnormalities) or unanticipated coronary revascularization, as positively adjudicated by the CEC.
Time Frame: From randomization to the first occurrence of any component of the composite secondary endpoint (median duration of follow-up was 39.9 months)
Population: All subjects randomized to treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dalcetrapib
Number analyzed (Participants) | 3076 | 3071
Participants | 471 | 471
Statistical Analysis 1: Comparison: Placebo vs Dalcetrapib; Secondary endpoints were expressed as time to event and an analysis similar to that for the primary endpoint was conducted. In order to control the family-wise Type I error that results from the multiplicity of endpoints, the secondary endpoints were formally tested using the Hochberg's step-up procedure only if the primary analysis results in significant treatment effect at p<0.05. Otherwise, statistical tests for the secondary endpoints were presented solely for illustrative purposes; Test type: Superiority; p = 0.95, Stratified Cox proportional hazard model; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.88 to 1.13]

3. Secondary Outcome: Composite Endpoint of Cardiovascular Death, Resuscitated Cardiac Arrest, Non-Fatal Myocardial Infarction, Non-Fatal Stroke or Hospitalization for New or Worsening Heart Failure
Description: All efficacy endpoints were adjudicated by an independent clinical endpoint committee (CEC). The secondary efficacy endpoint was the time from randomization to the first occurrence of any component of the composite secondary endpoint, which included death from cardiovascular causes, cardiovascular death, resuscitated cardiac arrest, non-fatal myocardial infarction, non-fatal stroke, or hospitalization for new or worsening heart failure, as positively adjudicated by the CEC.
Time Frame: as for outcome 2
Population: All subjects randomized to treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dalcetrapib
Number analyzed (Participants) | 3076 | 3071
Participants | 346 | 321
Statistical Analysis 1: Comparison: Placebo vs Dalcetrapib; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.27, Stratified Cox proportional hazard model; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.79 to 1.07]

ADVERSE EVENTS:
Time Frame: From randomization through 14 days after end of study (median duration of follow-up was 39.9 months).
Description: Positively adjudicated endpoints by the Clinical Endpoints Committee (CEC) as well as those negatively adjudicated by the CEC and reported as unrelated to study drug by the Investigators were exempted from SAE reporting.
  At each study visit after randomization the Investigator asked the patient if any untoward medical event occurred since the last visit. The date of onset and end, intensity, relationship to study medication, outcome, and treatments administered for the event(s) were recorded.
Arm/Group | Placebo | Dalcetrapib
All-Cause Mortality (participants affected / at risk) | 180/3076 | 182/3071
Serious Adverse Events (participants affected / at risk) | 923/3076 | 900/3071
Other Adverse Events (participants affected / at risk) | 818/3076 | 971/3071
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=3076) | Dalcetrapib (N=3071)
Anaemia (Blood and lymphatic system disorders) | 21 | 19
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Hemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 1
Hypchromic anaemia (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Non-Hodgkin's lymphoma recurrent (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Splenic haematoma (Blood and lymphatic system disorders) | 1 | 0
Splenic infarction (Blood and lymphatic system disorders) | 2 | 0
Splenic vein thrombosis (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Acute Coronary Syndrome (Cardiac disorders) | 0 | 1
Adams-Stokes Syndrome (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 50 | 52
Angina unstable (Cardiac disorders) | 23 | 19
Aortic valve disease (Cardiac disorders) | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 5 | 1
Arrhythmia (Cardiac disorders) | 3 | 2
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Arteriospasm coronary (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 36 | 31
Atrial flutter (Cardiac disorders) | 6 | 4
Atrial tachycardia (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 2 | 0
Atrioventricular block complete (Cardiac disorders) | 6 | 1
Atrioventricular block second degree (Cardiac disorders) | 3 | 4
Bradycardia (Cardiac disorders) | 3 | 7
Cardiac aneurysm (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 5 | 5
Cardiac failure (Cardiac disorders) | 4 | 7
Cardiac failure acute (Cardiac disorders) | 0 | 2
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cardiac valve disease (Cardiac disorders) | 0 | 1
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 2
Cardio-respiratory arrest (Cardiac disorders) | 2 | 4
Cardiogenic shock (Cardiac disorders) | 3 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 2
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0
Carditis (Cardiac disorders) | 0 | 1
Chest pain (Cardiac disorders) | 1 | 0
Cor pulmonale (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 23 | 30
Coronary artery dissection (Cardiac disorders) | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 3 | 2
Coronary artery perforation (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 7 | 7
Ischaemic cardiomyopathy (Cardiac disorders) | 2 | 3
Left ventricular dysfunction (Cardiac disorders) | 3 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0
Long QT syndrome (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 2
Myocardial haemorrhage (Cardiac disorders) | 1 | 0
Myocardia ischaemia (Cardiac disorders) | 12 | 12
Myocarditis (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 2 | 2
Pericardial effusion (Cardiac disorders) | 1 | 2
Pericarditis (Cardiac disorders) | 4 | 3
Right ventricular failure (Cardiac disorders) | 1 | 0
Sinus arrest (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 4 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 2
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 4 | 4
Systolic dysfunction (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 2 | 1
Ventricular fibrillation (Cardiac disorders) | 2 | 2
Ventricular tachycardia (Cardiac disorders) | 5 | 8
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0
Bicuspid aortic valve (Congenital, familial and genetic disorders) | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 3 | 0
Ear canal stenosis (Ear and labyrinth disorders) | 0 | 1
Meniere's disease (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 2
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0
Cushing's syndrome (Endocrine disorders) | 1 | 0
Hyperparathyroidism primary (Endocrine disorders) | 1 | 0
Thyroid mass (Endocrine disorders) | 1 | 0
Toxic goitre (Endocrine disorders) | 0 | 1
Blindness transient (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 1
Lens dislocation (Eye disorders) | 1 | 0
Optic nerve disorder (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 1 | 2
Retinal tear (Eye disorders) | 0 | 1
Retinopathy of prematurity (Eye disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 6 | 7
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 5 | 2
Adenocarcinoma pancreas (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Auriculotemporal syndrome (Gastrointestinal disorders) | 1 | 0
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 2
Coeliac artery stenosis (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 2 | 0
Colitis ischaemic (Gastrointestinal disorders) | 2 | 2
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 5
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Dysphagia (Gastrointestinal disorders) | 4 | 2
Enteritis (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 2 | 2
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 3 | 3
Gastritis erosive (Gastrointestinal disorders) | 1 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 8 | 5
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 4
Gingival recession (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 3
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 2
Hernial eventration (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 2 | 2
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Inflammatory bowel disease (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 5 | 5
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 3
Intestinal perforation (Gastrointestinal disorders) | 0 | 2
Large intestinal polyp (Gastrointestinal disorders) | 0 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 3
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 4 | 2
Mesenteric panniculitis (Gastrointestinal disorders) | 0 | 1
Oesophageal dysplasia (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 3 | 7
Pancreatitis acute (Gastrointestinal disorders) | 14 | 6
Pancreatitis chronic (Gastrointestinal disorders) | 3 | 1
Peptic ulcer (Gastrointestinal disorders) | 2 | 0
Portal venous gas (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 3
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 5
Small intestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 1
Umbilical hernia (Gastrointestinal disorders) | 2 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 2
Volvulus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 4
Asthenia (General disorders) | 2 | 3
Cardiac death (General disorders) | 1 | 0
Chest discomfort (General disorders) | 7 | 1
Chest pain (General disorders) | 79 | 81
Death of unknown cause (General disorders) | 8 | 17
Drowning (General disorders) | 1 | 0
Drug intolerance (General disorders) | 0 | 1
Exercise tolerance decreased (General disorders) | 2 | 0
Fatigue (General disorders) | 1 | 1
General physical health deterioration (General disorders) | 1 | 2
Generalized oedema (General disorders) | 0 | 1
Impaired self-care (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 1
Nodule (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 28 | 41
Oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Pacemaker generated arrhythmia (General disorders) | 1 | 0
Polyp (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 2
Sudden cardiac death (General disorders) | 3 | 8
Sudden death (General disorders) | 14 | 16
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Vascular stent restenosis (General disorders) | 3 | 2
Vascular stent stenosis (General disorders) | 1 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 2 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 2 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 2
Cholangitis acute (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 10 | 8
Cholecystitis acute (Hepatobiliary disorders) | 4 | 8
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 8 | 5
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Hepatic cyst (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1
Hepatic lesion (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 0 | 1
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 2
Drug hypersensitivity (Immune system disorders) | 0 | 1
Food allergy (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 2 | 1
Sarcoidosis (Immune system disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 2
Abscess limb (Infections and infestations) | 1 | 1
Abscess of salivary gland (Infections and infestations) | 0 | 1
Abscess oral (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 2 | 3
Appendicitis (Infections and infestations) | 8 | 7
Appendicitis perforated (Infections and infestations) | 1 | 0
Arteriosclerotic gangrene (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 2
Bacteraemia (Infections and infestations) | 1 | 1
Bacterial infection (Infections and infestations) | 0 | 1
Biliary sepsis (Infections and infestations) | 1 | 0
Brain abscess (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 4
Cardiac valve vegetation (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 12 | 12
Cellulitis staphylococcal (Infections and infestations) | 1 | 0
Central nervous system infection (Infections and infestations) | 1 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 2
Colonic abscess (Infections and infestations) | 0 | 1
Corona virus infection (Infections and infestations) | 43 | 45
Creutzfeldt-Jakob disease (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 3
Device related infection (Infections and infestations) | 1 | 0
Diabetic foot infection (Infections and infestations) | 0 | 2
Diarrhoea infectious (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 6 | 7
Ear infection (Infections and infestations) | 1 | 0
Eczema infected (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 2 | 0
Endocarditis bacterial (Infections and infestations) | 1 | 0
Epididymitis (Infections and infestations) | 2 | 1
Erysipelas (Infections and infestations) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Escherichia infection (Infections and infestations) | 0 | 1
Escherichia pyelonephritis (Infections and infestations) | 0 | 2
Gangrene (Infections and infestations) | 2 | 1
Gastric ulcer helicobacter (Infections and infestations) | 1 | 0
Gastritis bacterial (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 10 | 8
Gastroenteritis viral (Infections and infestations) | 4 | 4
Gastrointestinal infection (Infections and infestations) | 1 | 0
Haematoma infection (Infections and infestations) | 3 | 0
Haemophilus bacteraemia (Infections and infestations) | 1 | 0
Helicobacter infection (Infections and infestations) | 0 | 1
Hepatitis C (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 1
Herpes zoster oticus (Infections and infestations) | 0 | 1
Implant site infection (Infections and infestations) | 1 | 1
Infected lymphocele (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 1
Infectious colitis (Infections and infestations) | 0 | 1
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 3
Influenza (Infections and infestations) | 2 | 3
Klebsiella bacteraemia (Infections and infestations) | 2 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 2 | 2
Localized infection (Infections and infestations) | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 8 | 3
Lung abscess (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 1
Nosocomial infection (Infections and infestations) | 1 | 0
Ophthalmic herpes simplex (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 3 | 2
Osteomyelitis (Infections and infestations) | 4 | 3
Pancreas infection (Infections and infestations) | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 41 | 39
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia escherichia (Infections and infestations) | 1 | 0
Pneumonia legionella (Infections and infestations) | 0 | 1
Pneumonia necrotising (Infections and infestations) | 1 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Pneumonia viral (Infections and infestations) | 2 | 1
Postoperative wound infection (Infections and infestations) | 1 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 2
Pyelonephritis (Infections and infestations) | 2 | 7
Pyelonephritis acute (Infections and infestations) | 4 | 2
Pyelonephritis chronic (Infections and infestations) | 2 | 0
Respiratory syncytial viral infection (Infections and infestations) | 2 | 0
Respiratory tract infection (Infections and infestations) | 5 | 3
Respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Scrotal abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 19 | 14
Septic shock (Infections and infestations) | 8 | 10
Serratia bacteraemia (Infections and infestations) | 0 | 1
Shunt infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 3 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 1
Tracheobronchitis (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 7 | 17
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 8 | 3
Vestibular neuronitis (Infections and infestations) | 1 | 1
Viral infection (Infections and infestations) | 2 | 2
Wound infection (Infections and infestations) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Anastomotic complication (Injury, poisoning and procedural complications) | 1 | 0
Anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 4 | 3
Arterial bypass thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Arterial injury (Injury, poisoning and procedural complications) | 0 | 1
Arterial restenosis (Injury, poisoning and procedural complications) | 0 | 1
Bile duct stenosis traumatic (Injury, poisoning and procedural complications) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Chest injury (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 3
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 3 | 0
Costal cartilage fracture (Injury, poisoning and procedural complications) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 2
Electric shock (Injury, poisoning and procedural complications) | 1 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Eye burns (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 6 | 11
Femoral neck fracture (Injury, poisoning and procedural complications) | 4 | 0
Femur fracture (Injury, poisoning and procedural complications) | 6 | 5
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 2
Foreign body (Injury, poisoning and procedural complications) | 0 | 2
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1
Haematuria traumatic (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 3
Head injury (Injury, poisoning and procedural complications) | 2 | 2
Hip fracture (Injury, poisoning and procedural complications) | 1 | 4
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 3
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Incomplete spinal fusion (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 2 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 4
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 3 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 2
Meniscus injury (Injury, poisoning and procedural complications) | 2 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 2
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 2 | 0
Perirenal haematoma (Injury, poisoning and procedural complications) | 1 | 0
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Pst procedural discomfort (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 2
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 2 | 4
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 5
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 2
Snake bite (Injury, poisoning and procedural complications) | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 3 | 1
Stab wound (Injury, poisoning and procedural complications) | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 3 | 2
Subdural haemorrhage (Injury, poisoning and procedural complications) | 2 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 4 | 4
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 2
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft stenosis (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Vascular psudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Wound secretion (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Angiogram (Investigations) | 0 | 1
Arteriogram coronary (Investigations) | 1 | 4
Biopsy prostate (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 2 | 0
Blood folate decreased (Investigations) | 0 | 1
Blood potassium increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 0 | 1
Cardiac murmur (Investigations) | 0 | 1
Cardiac stress test abnormal (Investigations) | 0 | 1
Carotid bruit (Investigations) | 1 | 0
Catheterization cardiac (Investigations) | 1 | 0
Catheterisation cardiac abnormal (Investigations) | 1 | 0
Cystoscopy (Investigations) | 0 | 1
Diagnostic procedure (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 3 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Fibrin D dimer increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 2 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1
Occult blood positive (Investigations) | 1 | 0
Pancreatic enzymes increased (Investigations) | 1 | 0
Sleep study (Investigations) | 1 | 0
Staphylococcus test positive (Investigations) | 1 | 0
Stress echocardiogram abnormal (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 1
Utereroscopy (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Adult failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 6 | 3
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 3
Diabetes with hyperosmolarity (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 2
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 4
Hyperosmolar hyperglycemic state (Metabolism and nutrition disorders) | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Obesity (Metabolism and nutrition disorders) | 1 | 2
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 3
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 4
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 6
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Knee impingement syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Limb deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 4
Mobility decreased (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 9 | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 27 | 23
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 5
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 4
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 2
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 2 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 7
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 | 2
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 1 | 0
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 3
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Atypical fibroxanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign neoplasm of prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 3
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 6
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chest wall tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia stage 1 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 4
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Epstein-Barr virus associated lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Giant cell tumour of tendon sheath (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Hepatic cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intestina adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Laryngeal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 6
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oropharyngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 3
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Plasma cell myeloma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pleural neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 27 | 10
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Tongue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ureteral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Balance disorder (Nervous system disorders) | 2 | 0
Burning sensation (Nervous system disorders) | 0 | 1
Carotid artery disease (Nervous system disorders) | 1 | 1
Carotid artery occlusion (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 5 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1
Cauda equina syndrome (Nervous system disorders) | 2 | 0
Cerebral artery stenosis (Nervous system disorders) | 0 | 1
Cerebral haematoma (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 2
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Cervical radiculopathy (Nervous system disorders) | 1 | 1
Cervicobrachial syndrome (Nervous system disorders) | 1 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0
Coma (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 1 | 0
Dementia Alzheimer's type (Nervous system disorders) | 0 | 2
Diabetic ketoacidotic hyperglycaemic coma (Nervous system disorders) | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 8 | 3
Encephalopathy (Nervous system disorders) | 2 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Generalized tonic-clonic seizure (Nervous system disorders) | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 5
Hemiparesis (Nervous system disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 2 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Hypoglycaemic coma (Nervous system disorders) | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 2 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Lumbosacral radicuopathy (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 2 | 2
Monoparesis (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 1 | 1
Presyncope (Nervous system disorders) | 3 | 2
Radicular pain (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 2
Seizure (Nervous system disorders) | 3 | 1
Status epilepticus (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 28 | 24
Transient ischemic attack (Nervous system disorders) | 10 | 6
Tremor (Nervous system disorders) | 1 | 0
Vascular dementia (Nervous system disorders) | 0 | 1
Vertebral artery stenosis (Nervous system disorders) | 0 | 2
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1
Device dislocation (Product Issues) | 1 | 1
Device material issue (Product Issues) | 1 | 0
Alcohol abuse (Psychiatric disorders) | 1 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 1
Alcoholism (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1
Aphasia (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 5 | 3
Conversion disorder (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 3 | 2
Hallucinations, mixed (Psychiatric disorders) | 1 | 0
Mania (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1
Schizoaffective disorder (Psychiatric disorders) | 1 | 0
Somatic symptom disorder (Psychiatric disorders) | 1 | 0
Substance abuse (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 20 | 18
Anuria (Renal and urinary disorders) | 1 | 0
Bladder dysplasia (Renal and urinary disorders) | 0 | 1
Calculus bladder (Renal and urinary disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 2 | 0
Chronic kidney disease (Renal and urinary disorders) | 3 | 3
Haematuria (Renal and urinary disorders) | 9 | 13
Haemorrhage urinary tract (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 2
Micturition disorder (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 7
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 3 | 3
Renal failure (Renal and urinary disorders) | 0 | 4
Renal impairment (Renal and urinary disorders) | 1 | 3
Renal injury (Renal and urinary disorders) | 0 | 1
Renal pain (Renal and urinary disorders) | 0 | 1
Ureteric stenosis (Renal and urinary disorders) | 2 | 1
Ureterolithiasis (Renal and urinary disorders) | 1 | 5
Urethral haemorrhage (Renal and urinary disorders) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 4 | 9
Urinary tract infection (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 5 | 9
Breast cyst (Reproductive system and breast disorders) | 0 | 1
Breast disorder (Reproductive system and breast disorders) | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 1 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bullous lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 19 | 15
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 16
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal granuloma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Non-cardiogenic pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 8
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Xanthelasma (Skin and subcutaneous tissue disorders) | 0 | 1
Alcohol use (Social circumstances) | 0 | 1
Sight disability (Social circumstances) | 0 | 1
Aneurysm repair (Surgical and medical procedures) | 1 | 0
Angioplasty (Surgical and medical procedures) | 1 | 0
Arthrodesis (Surgical and medical procedures) | 0 | 1
Atherectomy (Surgical and medical procedures) | 0 | 1
Blood pressure management (Surgical and medical procedures) | 0 | 1
Bone lesion excision (Surgical and medical procedures) | 0 | 1
Cardiac ablation (Surgical and medical procedures) | 2 | 0
Cardiac pacemaker insertion (Surgical and medical procedures) | 3 | 1
Cardiac pacemaker replacement (Surgical and medical procedures) | 1 | 1
Cardiac rehabilitation therapy (Surgical and medical procedures) | 1 | 0
Cardiac resynchronisation therapy (Surgical and medical procedures) | 1 | 0
Cataract operation (Surgical and medical procedures) | 1 | 0
Cholecystectomy (Surgical and medical procedures) | 2 | 1
Cholelithotomy (Surgical and medical procedures) | 0 | 1
Colostomy closure (Surgical and medical procedures) | 0 | 1
Coronary angioplasty (Surgical and medical procedures) | 1 | 0
Coronary arterial stent insertion (Surgical and medical procedures) | 0 | 1
Coronary artery bypass (Surgical and medical procedures) | 1 | 1
Coronary revascularisation (Surgical and medical procedures) | 0 | 2
Finger amputation (Surgical and medical procedures) | 0 | 1
Gastrectomy (Surgical and medical procedures) | 1 | 0
Heart transplant (Surgical and medical procedures) | 1 | 1
Hepatectomy (Surgical and medical procedures) | 0 | 1
Hernia repair (Surgical and medical procedures) | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 3 | 1
Implantable defibrillator insertion (Surgical and medical procedures) | 11 | 2
Insertion of ambulatory peritoneal catheter (Surgical and medical procedures) | 0 | 1
Keratoplasty (Surgical and medical procedures) | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 0 | 1
Left atrial appendage occlusion (Surgical and medical procedures) | 0 | 1
Limb amputation (Surgical and medical procedures) | 1 | 1
Lithotripsy (Surgical and medical procedures) | 0 | 1
Medical device change (Surgical and medical procedures) | 0 | 1
Ophthalmic fluid drainage (Surgical and medical procedures) | 0 | 1
Ossiculoplasty (Surgical and medical procedures) | 1 | 0
Percutaneous coronary intervention (Surgical and medical procedures) | 0 | 2
Rehabilitation therapy (Surgical and medical procedures) | 1 | 0
Renal transpant (Surgical and medical procedures) | 0 | 1
Soft tissue flap operation (Surgical and medical procedures) | 0 | 1
Stem cell transplant (Surgical and medical procedures) | 1 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 0
Tumour excision (Surgical and medical procedures) | 1 | 0
Urethral dilation procedure (Surgical and medical procedures) | 0 | 1
Vascular graft (Surgical and medical procedures) | 0 | 1
Vitrectomy (Surgical and medical procedures) | 1 | 0
Accelerated hypertension (Vascular disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 5 | 4
Aortic aneurysm rupture (Vascular disorders) | 0 | 2
Aortic dissection (Vascular disorders) | 0 | 2
Aortic intramural haematoma (Vascular disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 9 | 4
Arterial insufficiency (Vascular disorders) | 0 | 1
Arterial occlusive disease (Vascular disorders) | 0 | 1
Arterial perforation (Vascular disorders) | 1 | 0
Arterial stenosis (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0
Arteritis (Vascular disorders) | 0 | 1
Blood pressure inadequately controlled (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 4
Embolism arterial (Vascular disorders) | 0 | 1
Embolism venous (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 10 | 7
Hypertensive crisis (Vascular disorders) | 5 | 6
Hypertensive emergency (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 7 | 7
Hypovolaemic shock (Vascular disorders) | 1 | 0
Intermittent claudication (Vascular disorders) | 3 | 3
Internal haemorrhage (Vascular disorders) | 0 | 1
Ischaemia (Vascular disorders) | 2 | 1
Lymphocele (Vascular disorders) | 0 | 1
Malignant hypertension (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 2 | 5
Peripheral arterial occlusive disease (Vascular disorders) | 5 | 7
Peripheral artery aneurysm (Vascular disorders) | 2 | 2
Peripheral artery occlusion (Vascular disorders) | 3 | 2
Peripheral artery stenosis (Vascular disorders) | 4 | 1
Peripheral embolism (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 5 | 4
Peripheral vascular disorder (Vascular disorders) | 2 | 7
Phlebitis (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0
Thromboangiitis obliterans (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
Varicose vein (Vascular disorders) | 1 | 0
Vasculitis (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=3076) | Dalcetrapib (N=3071)
Hypertension (Vascular disorders) | 266 | 277
Chest pain (General disorders) | 239 | 268
Diarrhoea (Gastrointestinal disorders) | 186 | 300
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 155 | 152

LIMITATIONS AND CAVEATS:
The main limitation of this study is the occurrence of the COVID-19 pandemic during study conduct.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/39/NCT02525939/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/39/NCT02525939/SAP_001.pdf